CLINICAL TRIAL: NCT05162846
Title: Methods for Increasing Genetic Testing Uptake in Michigan
Acronym: MiGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UMCC 2021.076; U01CA232827 (NIH); HUM00192898 (Other: University of Michigan)
Record Dates: First submitted 2021-12-08; First posted 2021-12-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Colorectal Cancer; Ovarian Cancer; Prostate Cancer; Pancreatic Cancer; Endometrial Cancer; History of Cancer
Keywords: Genetic testing; Genetic susceptibility to malignant neoplasm
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms; Endometrial Neoplasms | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Usual care (UC) (Active Comparator): Participants are provided with a link to the Michigan Department of Health and Human Services (MDHHS) informational website and are instructed to follow up with their oncology provider about genetic testing.
  Interventions: Other: Publicly available genetic testing resources
- Arm 2 - Virtual genetics navigator (Experimental): Participants receive access to an online genetics tool, the virtual genetics navigator, to help learn why and how to seek out genetic testing for hereditary cancer syndromes.
  Interventions: Behavioral: Virtual genetics navigator
- Arm 3 - Motivational interviewing (MI) (Experimental): Participants receive up to 2 phone calls from trained genetics health coaches who provide information about genetic testing and use motivational interviewing to encourage participants to seek out clinical genetic testing.
  Interventions: Behavioral: Motivational interviewing (MI)

INTERVENTIONS:
Other: Publicly available genetic testing resources — Participants may view the publicly available Michigan Department of Health and Human Services (MDHHS) website as they wish.
  Arms: Arm 1 - Usual care (UC)
Behavioral: Virtual genetics navigator — A mobile-optimized website/online genetic tool developed by investigators from the University of Michigan's Center for Health Communications Research (CHCR).
  Arms: Arm 2 - Virtual genetics navigator
Behavioral: Motivational interviewing (MI) — At least 2 phone calls delivered by trained genetic health coaches using motivational interviewing and providing genetic testing information.
  Arms: Arm 3 - Motivational interviewing (MI)

SUMMARY:
The primary purpose of this study is to compare three interventions, two experimental and one standard of care (usual care), to see if the experimental interventions will increase the likelihood of a participant obtaining guideline-concordant genetic testing. Eligible participants will be randomized (assigned) to one of the following interventions: 1) Virtual genetics navigator, a mobile-optimized website, designed by the investigators, that delivers tailored messages and content; 2) two motivational interviewing (MI) telephone calls delivered by trained genetics health coaches; or 3) usual care.

DETAILED DESCRIPTION:
This trial will be conducted in partnership with the Michigan Department of Health and Human Services (MDHHS) and a network of oncology practices in Michigan, the Michigan Oncology Quality Consortium (MOQC).

As of April 2023 we were approved by our IRB to expand our inclusion criteria and recruitment cohort. This expansion will enhance our reach to individuals who are not in the acute stages of clinical care as well as individuals who are not in oncology care currently yet still qualify for genetic testing based on their family history of cancer alone or in combination with any personal cancer history. These expansions will also support the unburdening of oncology practices - who continue to face downstream, resource-limiting affects from the COVID-19 pandemic - across the state. The goal and aims of the study remain the same.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English
* Access to the internet
* Completed the Family Health History Tool (FHHT)
* Meeting clinical criteria for genetic evaluation due to any of the below:

  1. Personal history of Breast cancer either:

     * i. Diagnosed under 50
     * ii. Personal or family history of triple negative breast cancer
     * iii. Ashkenazi Jewish ancestry
     * iv. Male proband
     * v. 1st or 2nd degree relative with ovarian cancer, pancreatic cancer, breast cancer diagnosed under 50, or male breast cancer
  2. Personal history of prostate cancer either:

     * i. Diagnosed under 50
     * ii. Ashkenazi Jewish ancestry
     * iii. 1st or 2nd degree relative with ovarian cancer, pancreatic cancer, breast cancer diagnosed under 50, or male breast cancer
  3. Personal history of any cancer or no personal history of cancer with either:

     * i. PREMM score ≥ 2.5%
     * ii. 1st degree relative with pancreatic, or male breast cancer
     * iii. 1st or 2nd degree relative with ovarian cancer
     * iv. 1st degree relative with any of these cancers diagnosed under 50: colon, endometrial, or breast
     * v. Ashkenazi Jewish ancestry and 1st or 2nd degree relative with breast cancer
  4. Personal history of endometrial cancer diagnosed under 50
  5. Personal history of colorectal cancer diagnosed under 50
  6. Personal history of renal cancer diagnosed under 46
  7. Personal history of sarcoma diagnosed under 46 and a 1st or 2nd degree relative with sarcoma, breast cancer, or brain cancer diagnosed under 56
  8. Personal history of brain cancer diagnosed under 46 and a 1st or 2nd degree relative with sarcoma, breast cancer, or brain cancer diagnosed under 56
  9. Personal history of any two of the following cancers with at least one of them diagnosed under 46: breast, sarcoma, or brain
  10. Personal history of ovarian cancer
  11. Personal history of pancreatic cancer
  12. Personal history of adrenal cortical carcinoma

Exclusion Criteria:

* Prior clinical germline genetic testing for cancer or already have an upcoming appointment scheduled with a genetics provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 831 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2025-07-13 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who complete clinical genetic testing at six months after randomization | 6 months after enrollment/randomization
  The primary outcome is completion of genetic testing (yes/no) at 6 months after randomization by patient self-report.

SECONDARY OUTCOMES:
Barriers to genetic testing, for participants who completed genetic testing | 6 months and 12 months after enrollment/randomization
  Participants who have completed genetic testing (before the 6- or 12-month time point for this survey) will be asked to respond to this 7-item, study-specific survey, developed by the investigators to assess the importance of specific barriers that were identified in a previous, observational study. Each item is scored on a scale from 1-5 (1=not at all; 5=extremely). The mean score for each question, across all participants who completed genetic testing, will be calculated in order to rank the barriers in importance. A higher mean score indicates greater importance of that specific barrier.
Barriers to genetic testing, for participants who did not yet complete genetic testing | 6 months and 12 months after enrollment/randomization
  Participants who have not yet completed genetic testing (before the 6- or 12-month time point for this survey) will be asked to respond to this 23-item, study-specific survey, developed by the investigators to assess the importance of specific barriers that were identified in a previous, observational study. Each item is scored on a scale from 1-5 (1=not at all, 5=strongly agree). The mean score for each question, across all participants who have not yet completed genetic testing, will be calculated in order to rank the barriers in importance. A higher mean score indicates greater importance of that specific barrier.
Motivators of genetic testing, for participants who completed genetic testing | 6 months and 12 months after enrollment/randomization
  Participants who have completed genetic testing (before the 6- or 12-month time point for this survey) will be asked to respond to this 5-item, study-specific survey, developed by the investigators to assess the importance of specific motivators for future testing. Each item is scored on a scale from 1-5 (1=not at all; 5=extremely). The mean score for each question, across all participants who completed genetic testing, will be calculated in order to rank the motivators in importance. A higher mean score indicates greater importance of that specific motivator.
Motivators of genetic testing, for participants who did not yet complete genetic testing | 6 months and 12 months after enrollment/randomization
  Participants who have not yet completed genetic testing (before the 6- or 12-month time point for this survey) will be asked to respond to this 5-item, study-specific survey, developed by the investigators to assess the importance of specific motivators for future testing. Each item is scored on a scale from 1-5 (1=not at all, 5=strongly agree). The mean score for each question, across all participants who have not yet completed genetic testing, will be calculated in order to rank the motivators in importance. A higher mean score indicates greater importance of that specific motivator.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Stoffel, MD, MPH, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerido LH, Griggs JJ, Resnicow K, Kidwell KM, Delacroix E, Austin S, Hanson EN, Bacon E, Koeppe E, Goodall S, Demerath M, Rizzo EA, Weiner S, Hawley ST, Uhlmann WR, Roberts JS, Stoffel EM. The Michigan Genetic Hereditary Testing (MiGHT) study's innovative approaches to promote uptake of clinical genetic testing among cancer patients: a study protocol for a 3-arm randomized controlled trial. Trials. 2023 Feb 10;24(1):105. doi: 10.1186/s13063-023-07125-2. PMID 36765432

DOCUMENTS (1):
  • Informed Consent Form (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT05162846/ICF_000.pdf